CLINICAL TRIAL: NCT03894774
Title: Evaluation of an Intensive Inpatient Psychotherapy Treatment for Severely and Early Traumatized Children - Clinical Pilot Study Including Multimodal Mri (MOSES)
Brief Title: Evaluation of an Intensive Inpatient Psychotherapy Treatment for Severely and Early Traumatized Children (MOSES)
Acronym: MOSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Collaborators: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Principal Investigator, Karl H Brisch, Head of the Department of Pediatric Psychosomatic Medicin and Psychotherapy, LMU Klinikum
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MOSES
Record Dates: First submitted 2018-12-19; First posted 2019-03-29 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Chronic Post-Traumatic Stress Disorder; Neuroses, Posttraumatic; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study was conducted in the following randomized waiting control design:
  After being included in the study at time T0 the children stay in Treatment-As-Usual (TAU) for at least three months and are then randomly assigned to the Intensive Inpatient Psychotherapy Treatment Group (IG) or the Waiting Control Group (WCG) after this TAU time period (This period is considered necessary and sufficient in order to reliably estimate possible trends of changes in the brain). The children in the WCG stay in TAU and are assigned to the IG as soon as a treatment place is available. The waiting period will be included in the analysis as a confounder. The third group is a Healthy Control Group (HCG) of matched pairs (matched for gender, age and handedness).
Who Masked: Outcomes Assessor
Masking Description: Pseudonymization at first stage of the intervention. Additional anonymization for all outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intensive InPatient Psychotherapy Treatment Group (IG) (Experimental): Intensive non-pharmaceutical inpatient intervention with high degrees of individual psychotherapy (5 sessions a week, psychodynamic and specific trauma therapy), group therapy (music-, arts-, sports- and concentrative movement therapy - each one session a week) as well as an ongoing milieutherapeutic frame where patients live over the whole treatment (approximately a 1:1-ratio caregiver per patient is given) of 6 to 8 month treatment duration.
  Interventions: Behavioral: Intensive in-patient psychotherapy treatment
- Waiting Control Group (WCG) (Active Comparator): Treatment as usual (mostly combination of behavioral or psychoanalytic outpatient psychotherapy and pharmacotherapy).
  Duration: At least 3 month to a maximum of 6 month.
  Interventions: Other: Treatment as usual
- Healthy Control Group (HCG) (No Intervention): Matched Pairs design to control for gender, age and handedness. HCG measurements are planned and conducted according to the exact durations of their matched inpatient pair of the IG.
  Mandatory to control for effects of factors such as brain maturation.

INTERVENTIONS:
Behavioral: Intensive in-patient psychotherapy treatment — Intensive non-pharmaceutical in-patient intervention with high degrees of individual psychotherapy (5 sessions a week, psychodynamic and specific trauma therapy), group therapy (music-, arts-, sports- and concentrative movement therapy - each one session a week) as well as an ongoing milieutherapeutic setting where patients live during the whole treatment (approximately a 1:1-Ratio caregiver per patient is given) of 6 to 8 month treatment duration.
  Arms: Intensive InPatient Psychotherapy Treatment Group (IG)
Other: Treatment as usual — Combination of behavioral or psychoanalytic outpatient psychotherapy and pharmacotherapy
  Arms: Waiting Control Group (WCG)

SUMMARY:
Evaluation of longitudinal treatment effects applying an intensive psychotherapeutic intervention for inpatients (age of participants: 6-13 years) with a multi-method-approach to address the complex nature of severe childhood trauma. (Chronic Post-Traumatic Stress Disorder)

DETAILED DESCRIPTION:
Severe adversity and trauma in early childhood have been associated with a highly increased risk for a variety of psychiatric disorders, lasting into adulthood. This increased risk is accompanied by a set of biological changes ranging from changes in cortical thickness to endocrinological changes. At a behavioral level, children with complex PTSD (developmental trauma disorder) show severe and long-lasting negative effects. Such children exhibit a wide range of symptoms: affect dysregulation, attention difficulties, impairment in interpersonal relationships, aggressive and dissociative behaviour, disturbances of cognition. Corresponding alterations in neural networking and brain development are well studied. Although evidence-based treatment approaches for children with non-complex PTSD exist, complex-traumatized children have no well-evaluated treatments. Furthermore, early intervention can prevent the chronification and exacerbation of symptoms and promote social adaptation and participation.The following topics will be addressed: (1) brain development (Multimodal MRI (mMRI) including anatomical (T1-MPRAGE, T2-FLAIR, DTI-Diffusion Tensor Imaging) and functional MRI measurements (resting-state functional MRI, task fMRI (presenting affective pictures according to the International Affective Picture System, IAPS), EEG); (2) alterations in neuroendocrinological systems involved in stress regulation (Cortisol, Oxytocin, Vasopressin); (3) behavioral symptoms; (4) cognitive functioning; (5) attachment representations of children and their primary caregivers;

ELIGIBILITY:
Inclusion Criteria:

* Severe early traumatization with experiences of violence, neglect, abuse and chronic symptoms related to complex PTSD.

Exclusion Criteria:

* Autism spectrum disorder
* Addiction disorder
* Mental disability (IQ < 85)
* Endangerment to themselves or others

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Structural MRI (T1w, T2w, DTI) | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  All structural images will be acquired in a 3 Tesla MR system using a 20- channel head-coil (Siemens, Erlangen). Data post-processing will be performed with lab-internal scripts developed for a multi-core cluster. For structural analyses of T1w, T2w and DTI data, freesurfer,FSL and workbench will be used. T1w and T2w data will be volumetrically analyzed and the results will be reported in mm3. DTI data will be processed using tbss-FSL and probtrackX-FSL. DTI will be quantified in regard of the number of white matter fiber bundles within regions-of-interest (ROIs) and from-ROI-to-ROI. The Dosenbach atlas (Dosenbach et al. 2010) and the multimodal Brainetome atlas (Fan et al. 2016) will be used for all structural analyses. It is an explorative study that follows a whole-brain approach. Changes in emotion-processing and trauma-associated brain regions such as the hippocampus,the amygdala,the orbitofrontal cortex and the insula are assumed
Resting state functional MRI connectivity (rsfcMRI) | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  EPI-sequence: fMRI will be carried out at 3 Tesla (Siemens) scanner using a 20- channel head-coil. For functional imaging, an EPI sequence with the following parameters will be used: repetition time (TR),2000 ms; echo time (TE),30 ms; flip angle (FA), 80°; spatial resolution, 3 × 3 × 3 mm3; imaging matrix, 64 × 64; field-of-view (FoV), 192 × 192 mm2; number of slices: 36; number of volumes: 200. Data post-processing will be performed with lab-internal scripts developed for a multicore cluster. For rsfcMRI analyses of freesurfer,FSL,AFNI and workbench will be used. rsfcMRI will be quantified as number of significant activated voxels (spatial extent) and connectivity strength (z-scores).Networks of interest (ICA-based): Salience network, Default Mode Network. Regions of interest (seed-based): hippocampus, the amygdala, the orbitofrontal cortex and the insula.In addition, a RS-EEG with 19 scalp electrodes is used to complement rsfcMRI,which is cortically evaluated using Brainstorm.
Task-based fMRI using the International affective picture system (IAPS) | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  For the task-based fMRI the same EPI sequence will be used as for the resting state (see outcome 2). The number of volumes: 180. Three different sets of each 45 (15 neutral, 15 negative, 15 positive rated pictures) pictures were created and randomly displayed during the scanning procedure and also afterward to control for personal affective valence and arousal with Self-Assessment Manikin (SAM).
  Data post-processing will be performed with FSL-FEAT using a block-design. Regions of interest follow the previous structural and rsfcMRI analyses ROIs: hippocampus, amygdala, orbitofrontal cortex and the insula.

SECONDARY OUTCOMES:
Alterations in neuroendocrinological systems involved in stress regulation | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Oxytocin (pg/ml in Saliva) release of active stress regulation throughout relaxation using attachment interviews as stressors. Oxytocin will be analysed using radioimmunoassays in an external lab (Landgraf Riagnosis, MPI).
Alterations in neuroendocrinological systems involved in stress regulation 2 | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Cortisol (ng/mL in Saliva) release in active stress regulation throughout relaxation using attachment interviews as stressors. Cortisol will be analysed by Endocrine Laboratories, Department of Medicine IV, University Hospital, LMU Munich.
Alterations in neuroendocrinological systems involved in stress regulation 3 | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Vasopressin (pg/ml in Saliva) release of active stress regulation throughout relaxation using attachment interviews as stressors. Vasopressin will be analysed using radioimmunoassays in an external lab (Landgraf Riagnosis, MPI).

OTHER OUTCOMES:
Behavioral Symptoms 1: Child Behaviour Checklist (CBCL) | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Total Problems Score: 0-28="normal", 29-37="borderline", 38-236="clinical"
Behavioral Symptoms 2: Child Behaviour Checklist (CBCL) | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Externalizing Behaviour: 0-12="normal", 13-16="borderline", 17-66="clinical";
Behavioral Symptoms 3: Child Behaviour Checklist (CBCL) | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Internalizing Behaviour: 0-7="normal", 8-9="borderline", 10-62="clinical";
Behavioral Symptoms 4: Strength and Difficulties Questionnaire (SDQ). | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Total difficulties score: 0-13="normal", 14-16="borderline", 17-40="abnormal";
Behavioral Symptoms 5: Strength and Difficulties Questionnaire (SDQ). | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  hyperactivity score: 0-5="normal", 6="borderline", 7-10="abnormal"
Posttraumatic Symptoms | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Parent Repot of Posttraumatic Symptoms (PROPS). If total testscore is greater than 16 a posttraumatic stress disorder is suspected. Total Score range: 0-60.
Dissociation Symptoms | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Child Dissociation Scale (CDC). If total testscore is greater than 11 a dissociative disorder is suspected. Total Score range: 0-18.
Depression Symptoms | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Depression Inventory for Children and Young People (DIKJ - Depressionsinventar für Kinder und Jugendliche) If the testscore is greater than 14 a depression is suspected. Testscore range: 0-58.
Anxiety Symptoms | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Anxiety Questionnaire (FAS - Fragebogen für Angststörungen). If total testscore is greater than 24 a anxiety disorder is suspected. Total testscore range 0-82.
Cognitive Functioning | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Working Memory form Wechsler Intelligence Scale for Children (WISC-IV).
  At t0/t1 a full-scale intelligence test was conducted (IQ). To minimize learning effects through rehearsal, we focused on subtests in the follow-up testing:
  1. Digit Span (forward, backward)
  2. Letter-Number Sequencing
  By combining both subtest scores we calculate the Working Memory Index Score. The Working Memory Index will be used to address changes in cognitive functioning.
Attachment Representations | longitudinal (4 measurements, t0: at least 3 month before treatment, t1: at admission to treatment, t2: at discharge (average of 8 month), t3: 6 month post treatment)
  Child Attachment Interview (CAI). Changes in attachment representations in a qualitative binary secure-insecure distinction and in a four category qualitative coding classification (secure, dismissing, preoccupied, disorganized).

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Ebeling, M.A., Principal Investigator — Department of Pediatrics, Dr. von Hauner Children's Hospital, University Hospital, LMU Munich; Catherina Dehmel, M.sc., Principal Investigator — Department of Pediatrics, Dr. von Hauner Children's Hospital, University Hospital, LMU Munich; Lukas Oberschneider, MD, Principal Investigator — Department of Pediatrics, Dr. von Hauner Children's Hospital, University Hospital, LMU Munich
Locations (1):
- Department of Pediatrics, Dr. von Hauner Children's Hospital, University Hospital, LMU Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD concerning MRI analysis. Individual participant data set.
Supporting Information: Study Protocol, Analytic Code
Time Frame: 2019-2020
Access Criteria: MRI analyses

REFERENCES:
- [Background] Heim C, Binder EB. Current research trends in early life stress and depression: review of human studies on sensitive periods, gene-environment interactions, and epigenetics. Exp Neurol. 2012 Jan;233(1):102-11. doi: 10.1016/j.expneurol.2011.10.032. Epub 2011 Nov 7. PMID 22101006
- [Background] Hamilton, L., Micol-Foster, V., & Muzik, M. Childhood maltreatment trauma: Relevance for adult physical and emotional health. A Review. Trauma Cases and Reviews, 1(003), 2015.
- [Background] D'Andrea W, Ford J, Stolbach B, Spinazzola J, van der Kolk BA. Understanding interpersonal trauma in children: why we need a developmentally appropriate trauma diagnosis. Am J Orthopsychiatry. 2012 Apr;82(2):187-200. doi: 10.1111/j.1939-0025.2012.01154.x. PMID 22506521
- [Background] Pechtel P, Pizzagalli DA. Effects of early life stress on cognitive and affective function: an integrated review of human literature. Psychopharmacology (Berl). 2011 Mar;214(1):55-70. doi: 10.1007/s00213-010-2009-2. Epub 2010 Sep 24. PMID 20865251
- [Background] Teicher MH, Samson JA, Anderson CM, Ohashi K. The effects of childhood maltreatment on brain structure, function and connectivity. Nat Rev Neurosci. 2016 Sep 19;17(10):652-66. doi: 10.1038/nrn.2016.111. PMID 27640984
- [Background] Gold AL, Sheridan MA, Peverill M, Busso DS, Lambert HK, Alves S, Pine DS, McLaughlin KA. Childhood abuse and reduced cortical thickness in brain regions involved in emotional processing. J Child Psychol Psychiatry. 2016 Oct;57(10):1154-64. doi: 10.1111/jcpp.12630. PMID 27647051
- [Background] Gillies D, Taylor F, Gray C, O'Brien L, D'Abrew N. Psychological therapies for the treatment of post-traumatic stress disorder in children and adolescents (Review). Evid Based Child Health. 2013 May;8(3):1004-116. doi: 10.1002/ebch.1916. PMID 23877914